CLINICAL TRIAL: NCT05705674
Title: The Natural History Study of Patients With Sanfilippo Disease(s) (MPS3)
Status: Recruiting | Type: Observational
Sponsor: Lysosomal and Rare Disorders Research and Treatment Center, Inc. (Other)
Collaborators: Team Sanfilippo (Unknown)
Responsible Party: Sponsor
Other Study IDs: 22-LDRTC-01
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Sanfilippo Syndrome; MPS3
MeSH Terms: conditions — Mucopolysaccharidosis III

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The natural history study of patients with Sanfilippo disease(s) (MPS3)

DETAILED DESCRIPTION:
This is a natural history study of patients with Sanfilippo Disease (MPS3). Patients will be followed over the course of 6 months in which they have blood and urine collected, hearing assessment, complete questionnaires and are evaluated by the Principal Investigator.

ELIGIBILITY:
Inclusion Criteria:

1. IRB - approved informed consent/assent signed by subject and/or parent(s) or legal guardian(s).
2. Genetically confirmed diagnosis of MPS III disease Genomic DNA analysis demonstrating a homozygous or compound heterozygous pathogenic variants in SGSH (type A), NAGLU (type B), HGSNAT (type C), or N- acetylglucosamine-6-sulfatase GNS (type D).
3. Male or female; five years of age and older
4. Negative urine pregnancy test at screening for female subjects with child-bearing potential

Exclusion Criteria:

1. Unwilling or unable to follow protocol requirements as per principal investigator
2. Any serious or chronic medical illness, including significant cardiac or severe debilitating pulmonary disease as determined by the investigator.
3. Any medical condition that, in the opinion of the PI, would place a subject at undue risk
4. Inability to cooperate for clinical and safety data collection
5. Use of genistein or Miglustat within one week of the study
6. Evidence of hepatitis B or hepatitis C infection upon serological testing at screening
7. Currently participating in another interventional drug trial or has completed an interventional trial less than one month prior to the screening visit

Ages: 5 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with MPS3 who meet the criteria above can be enrolled.
Sampling Method: Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To characterize the disease natural history in patients with MPS3. | 6 months
  To characterize the disease natural history in patients with MPS3.

CONTACTS AND LOCATIONS:
Locations (1):
- LDRTC, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
No plan to make IPD available to other researchers.